CLINICAL TRIAL: NCT05236894
Title: Examining the Appeal of Nicotine Pouches in Ohio Appalachia
Brief Title: Appeal of Nicotine Pouches Versus Cigarettes in the Ohio Appalachia Population
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brittney Keller-Hamilton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-21257; NCI-2021-14062 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-01-13; First posted 2022-02-11 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — WD repeat containing planar cell polarity effector

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Aim 1: Arm I (lower dose nicotine pouch) (Experimental): Patients receive lower dose nicotine pouch PO over 30 minutes at visits 1, 2, and 3.
  Interventions: Drug: Nicotine Oral Pouch; Other: Questionnaire Administration
- Aim 1: Arm II (higher dose nicotine pouches) (Experimental): Patients receive higher dose nicotine pouch PO over 30 minutes at visits 1, 2, and 3.
  Interventions: Drug: Nicotine Oral Pouch; Other: Questionnaire Administration
- Aim 1: Arm III (cigarette smoking) (Active Comparator): Patients smoke usual brand of cigarettes, taking one puff every 30 seconds over 5 minutes at visits 1, 2, and 3.
  Interventions: Behavioral: Cigarette Smoking; Other: Questionnaire Administration
- Aim 2: Arm I (3mg NP) (Experimental): Patients receive nicotine pouch PO over 30 minutes at visits 1, 2, and 3.
  Interventions: Other: Questionnaire Administration; Drug: Nicotine Oral Pouch
- Aim 2: Arm II (3mg NP) (Experimental): Patients receive nicotine pouch PO over 30 minutes at visits 1, 2, and 3.
  Interventions: Other: Questionnaire Administration; Drug: Nicotine Oral Pouch
- Aim 2: Arm III (3mg NP) (Experimental): Patients receive nicotine pouch PO over 30 minutes at visits 1, 2, and 3.
  Interventions: Other: Questionnaire Administration; Drug: Nicotine Oral Pouch

INTERVENTIONS:
Behavioral: Cigarette Smoking — Smoke preferred brand of cigarette
  Arms: Aim 1: Arm III (cigarette smoking)
Drug: Nicotine Oral Pouch — Given lower dose nicotine pouch
  Other Names: ZYN
  Arms: Aim 1: Arm I (lower dose nicotine pouch)
Drug: Nicotine Oral Pouch — Given higher dose nicotine pouch
  Other Names: ZYN
  Arms: Aim 1: Arm II (higher dose nicotine pouches)
Other: Questionnaire Administration — Ancillary studies
Drug: Nicotine Oral Pouch — Given 3mg nicotine pouch (Aim 2)
  Other Names: On!
  Arms: Aim 2: Arm I (3mg NP)
Drug: Nicotine Oral Pouch — Given 3mg nicotine pouch (Aim 2)
  Other Names: ZYN
  Arms: Aim 2: Arm II (3mg NP)
Drug: Nicotine Oral Pouch — Given 3mg nicotine pouch (Aim 2)
  Other Names: Fre
  Arms: Aim 2: Arm III (3mg NP)

SUMMARY:
This clinical trial estimates the abuse liability of nicotine pouches with varying nicotine concentrations relative to cigarette smoking in Appalachian, Ohio and Ohio smokers. Nicotine pouches are a novel tobacco product with potential to reduce or increase the harm of tobacco use. Evaluating nicotine pouches abuse liability among smokers in Ohio including the unique demographic of Appalachia may clarify the public health effect of NPs in Appalachian Ohio and across Ohio. Results may inform public health efforts, policy, and clinical care aimed at reducing tobacco-related disparities.

DETAILED DESCRIPTION:
Aim 1:

PRIMARY OBJECTIVE:

I. To estimate the abuse liability of nicotine pouches (NPs) with varying nicotine concentrations relative to cigarette smoking.

SECONDARY OBJECTIVE:

I. To clarify the public health effect of NPs in Appalachian Ohio.

EXPLORATORY OBJECTIVES:

I. To estimate the abuse liability of NPs with varying nicotine concentrations relative to cigarette smoking by measuring nicotine pharmacokinetics.

II. To estimate the abuse liability of NPs with varying nicotine concentrations relative to cigarette smoking by measuring subjective effects.

III. To estimate the abuse liability of NPs with varying nicotine concentrations relative to cigarette smoking by measuring intentions to use and switch to NPs.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive lower dose nicotine pouch orally (PO) over 30 minutes at visits 1, 2, and 3.

ARM II: Patients receive higher dose nicotine pouch PO over 30 minutes at visits 1, 2, and 3.

ARM III: Patients smoke usual brand of cigarettes, taking one puff every 30 seconds over 5 minutes at visits 1, 2, and 3.

Aim 2:

PRIMARY OBJECTIVE:

I. To understand the pharmacokinetic difference between tobacco-derived and synthetic NPs.

SECONDARY OBJECTIVE:

I. To clarify the public health effect of NPs on adult smokers

EXPLORATORY OBJECTIVES:

I. To understand the differences in abuse liability between tobacco-derived and synthetic NPs by measuring nicotine pharmacokinetics.

II. To understand the differences in abuse liability between tobacco-derived and synthetic NPs by measuring subjective effects.

III. To estimate the abuse liability of tobacco-derived vs. synthetic NPs by measuring intentions to use and switch to NPs.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive a 3mg dose nicotine pouch orally (PO) over 30 minutes at visits 1, 2, and 3.

ARM II: Patients receive a 3mg dose nicotine pouch PO over 30 minutes at visits 1, 2, and 3.

ARM III: Patients receive a 3mg dose nicotine pouch PO over 30 minutes at visits 1, 2, and 3.

ELIGIBILITY:
Aim 1 Inclusion Criteria:

* Age 21 years or older.
* Reside in an Ohio Appalachian county.
* Willing to complete study procedures, including abstaining from all tobacco, nicotine, and marijuana for 12 hours before clinic visits.
* Ability to read and speak English.
* Smoke at least 5 cigarettes per day for the past 30 days.

Exclusion Criteria:

* Use tobacco products other than cigarettes >10 days per month.
* Use NP in the past 3 months.
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed).
* Pregnant, planning to become pregnant, or breastfeeding.
* History of cardiac event or distress within the past 3 months.
* Currently attempting to quit all tobacco use.
* Self-reported diagnosis of lung disease including asthma (if uncontrolled or worse than usual), cystic fibrosis, or chronic obstructive pulmonary disease.

Aim 2 Inclusion Criteria:

* Age 21 years or older.
* Reside in a Ohio.
* Willing to complete study procedures, including abstaining from all tobacco, nicotine, and marijuana for 12 hours before clinic visits.
* Ability to read and speak English.
* Smoke at least 5 cigarettes per day for the past 30 days.

Exclusion Criteria:

* Use tobacco products other than cigarettes >10 days per month.
* Use NP in the past 3 months.
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed).
* Pregnant, planning to become pregnant, or breastfeeding.
* History of cardiac event or distress within the past 3 months.
* Currently attempting to quit all tobacco use.
* Self-reported diagnosis of lung disease including asthma (if uncontrolled or worse than usual), cystic fibrosis, or chronic obstructive pulmonary disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Evaluate plasma nicotine concentration at t=30 minutes for each product. | Up to 6 months

SECONDARY OUTCOMES:
Aim 1: Public health effect of NPs in Appalachian Ohio - if NPs can be used as a substitute for cigarette smoking | Up to 6 months
  Data collected will show if NPs are a viable substitute for cigarette smoking.
Evaluate plasma nicotine concentrations at t=5 through t=90 minutes | Up to 6 months
Evaluate withdrawal relief at t=5 through t=90 minutes | Up to 6 months
  We measure withdrawal relief using the Minnesota Withdrawal Scale (MNWS). We administer this questionnaire at each timepoint along the standardized scale of t=0, t=5, t=15, t=30, t=60 and t=90. The MNWS includes a minimum value of "none" and a maximum value or "severe." The higher scores indicate increased withdrawal symptoms and lower scores indicate lessened or no withdrawal symptoms.
Evaluate product appeal across all 3 products | Up to 6 months
  Product appeal will be assessed using several scales, including the Modified E-Cigarette Smoking Questionnaire (mCEQ), the Product Evaluation Scale (PES), the Adapted Drug Effects Liking Scale, and the Study Product Effects Liking Scale which are administered after the final timepoint of each study visit. For both the mCEQ and PES, the minimum scale value is "not at all" and the maximum scale value is "extremely." Higher scores can mean both better or worse depending on the question. Ex: "Was using your smokeless tobacco satisfying?" and "Did using your smokeless tobacco make you nauseous?" are both questions on each scale, so a higher score would vary in meaning based on the question. For the Adapted Drug Effects Liking and Study Product Effects Liking scales, minimum values include "not at all" and maximum value includes "very pleasant." With the exception of one question on the Study Product Effects Liking Scale, a higher score indicates increased enjoyment of the product.

OTHER OUTCOMES:
Aim 1 and 2: Nicotine pharmacokinetics | Up to 6 months
  Will use linear or logistic mixed effects regression models (with a random subject effect) to assess the main effects of product on plasma nicotine delivery.
Subjective effects - likability and substitutability of product compared to cigarette smoking will be assessed | Up to 6 months
  Will use linear or logistic mixed effects regression models (with a random subject effect) to assess the main effects of product on subjective effects.
Aim 1: Intentions to use and switch to NPs - quit intentions will be assessed using a 10 question survey | Up to 6 months
  Will use linear or logistic mixed effects regression models (with a random subject effect) to assess the main effects of product behavioral intentions.
Aim 2: Public health effect of NPs in adult smokers - if NPs can be used as a substitute for cigarette smoking. | Up to 6 months
  Public health impact of NPs in adult smokers as an alternative for cigarette smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney L Keller-Hamilton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller-Hamilton B, Alalwan MA, Curran H, Hinton A, Long L, Chrzan K, Wagener TL, Atkinson L, Suraapaneni S, Mays D. Evaluating the effects of nicotine concentration on the appeal and nicotine delivery of oral nicotine pouches among rural and Appalachian adults who smoke cigarettes: A randomized cross-over study. Addiction. 2024 Mar;119(3):464-475. doi: 10.1111/add.16355. Epub 2023 Nov 14. PMID 37964431
- [Background] Keller-Hamilton B, Curran H, Alalwan M, Hinton A, Brinkman MC, El-Hellani A, Wagener TL, Chrzan K, Atkinson L, Suraapaneni S, Mays D. Evaluating the Role of Nicotine Stereoisomer on Nicotine Pouch Abuse Liability: A Randomized Crossover Trial. Nicotine Tob Res. 2025 Mar 24;27(4):658-665. doi: 10.1093/ntr/ntae079. PMID 38713545
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT05236894/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT05236894/ICF_001.pdf